CLINICAL TRIAL: NCT03285620
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, First-in-human Study of Orally Administered AL-034 to Evaluate the Safety, Tolerability, and Pharmacokinetics After Single Ascending Doses Including Food Effect Evaluation (Part 1) and After Multiple Ascending Doses (Part 2) in Healthy Adult Subjects
Brief Title: A Study of AL-034 to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AL-034-1201; AL-034-1201 (Other: Alios BioPharma Inc.)
Record Dates: First submitted 2017-08-15; First posted 2017-09-18 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Single Ascending Dose (SAD) (Experimental): Participants will receive single oral dose of AL-034 (oral solution) (the starting dose in Cohort 1 of Part 1 will be 0.2 milligram [mg]) or matching placebo under fasted condition (Cohorts 1 to 5 or optional Cohort 7) on Day 1. Participants may receive AL-034 in a fed state (Cohort 6) to evaluate the effect of food on the pharmacokinetics (PK) of AL-034.
  Interventions: Drug: AL-034; Drug: Placebo
- Part 2: Multiple-Dose Administration (MAD) (Experimental): Participants will receive multiple oral doses of AL-034 or matching placebo for 4 consecutive weeks either once weekly (Qwk - for 4 doses) or every two weeks (Q2wk - for 3 doses) under fed or fasted conditions. The starting dose for Part 2 will be determined based on the initial PK and safety/tolerability data from Part 1.
  Interventions: Drug: AL-034; Drug: Placebo

INTERVENTIONS:
Drug: AL-034 — Participants will receive single oral dose of AL-034 under fed or fasted conditions in part 1 and part 2
Drug: Placebo — Participants will receive single oral dose of matching placebo (oral solution) under fed or fasted conditions in part 1 and part 2.

SUMMARY:
This is a Phase 1 first-in-human (FIH) study evaluating single and multiple dose administration of AL-034 in healthy adult participants. The aim is to examine the safety (including pharmacodynamic [PD] biomarker assessments), tolerability, and pharmacokinetics (PK) of increasing single ascending doses (SADs) (Part 1) and multiple ascending doses (MADs) (Part 2) of AL-034. The potential food effect will be investigated in healthy adult participants at one or optionally 2 single dose level(s).

ELIGIBILITY:
INCLUSION CRITERIA Each potential participant must satisfy all of the following criteria to be enrolled in the study

* participant must be a man or a woman between 18 and 55 years of age, extremes included
* Female participant must be of non-childbearing potential, defined as: a) Postmenopausal: A postmenopausal state is defined as no menses for 12 months without an alternative medical explanation. A high follicle stimulating hormone (FSH) level (greater than [>]40 international unit per liter [IU/L] or milli international unit per milliliter [mIU/mL]) in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, 2 FSH measurements will have to be taken at least 3 months apart, OR b) Permanently sterile - permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy Male participants must either: a) be surgically sterile (have had a vasectomy), or otherwise incapable of fathering a child, OR b) if heterosexually active, have a partner who is postmenopausal (as defined above), permanently sterile (as defined above), or otherwise incapable of becoming pregnant, OR c) if heterosexually active with a woman of childbearing potential, agree to use effective methods of contraception as detailed in Prohibitions and Restrictions section, from screening onwards, and agree to continue to use the same method of contraception throughout the study and for at least 90 days after the last dose of study drug Contraceptive use should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies
* Female participants should have a negative pregnancy test at screening and on Day -1
* Participants must be non-smokers for at least 3 months prior to screening
* Participants must have a body mass index (BMI; weight in kilogram [kg] divided by the square of height in meters) of 18.0 to 30.0 kilogram per meter square (kg/m^2), extremes included. (Williamson 1993)
* Participants must have a normal 12-lead electrocardiogram (ECG) (based on the mean value of the triplicate parameters) at screening including: a) Normal sinus rhythm (heart rate between 50 and 100 beats per minute [bpm], extremes included); b) QT interval corrected for heart rate (QTc) according to Fridericia's formula (QTcF) less than or equal to (<=)450 millisecond (ms) (Fridericia 1920); c) QRS interval less than (<)120 ms; d) PR interval <=200 ms; e) ECG morphology consistent with healthy cardiac conduction and function. Any evidence of heart block is exclusionary. Any evidence of left or right bundle branch block is exclusionary Note: Retesting for abnormal QTc interval value that may lead to exclusion will be allowed once without prior approval from the Sponsor. Retesting may take place during an unscheduled visit in the screening phase. Participants with a normal value at retest may be included
* Participants must be healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, vital signs, and the results of blood chemistry, blood coagulation and hematology tests, and a urinalysis performed at screening
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in Prohibitions and Restrictions section
* In the Investigator's opinion, the participant is able to understand and comply with protocol requirements, instructions, and study restrictions and is likely to complete the study as planned
* Participant must sign a separate if he or she agrees to provide an optional deoxyribonucleic acid (DNA) sample for research. Refusal to give consent for the optional DNA research sample does not exclude a participant from participation in the study

EXCLUSION CRITERIA Any potential participant who meets any of the following criteria will be excluded from participating in the study

* Participants with a past history of cardiac arrhythmias (for example, extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (for example, hypokalemia, family history of long QT Syndrome) or history or other clinical evidence of significant or unstable cardiac disease (for example, angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia, coronary heart disease, and/or clinically significant ECG abnormalities), moderate to severe valvular disease or uncontrolled hypertension at screening. Any evidence of heart block or bundle branch block is also exclusionary
* Participants with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant or that could prevent, limit, or confound the protocol specified assessments. This may include but is not limited to renal dysfunction (estimated creatinine clearance below 60 milliliter per minute [mL/min] at screening, calculated by the Modification of Diet in Renal Disease [MDRD] formula [Poggio 2005]), significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the Investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, ophthalmic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances. Any condition possibly affecting drug absorption (for example, gastrectomy or other significant gastrointestinal tract surgery, such as gastroenterostomy, small bowel resection, or active enterostomy) will also lead to exclusion
* Participants with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria
* Participants with a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs
* Participants with a history or current evidence of use of alcohol, amphetamines, barbiturates, recreational or narcotic drug use within the past 1 year, which in the Investigator's opinion would compromise Participant's safety and/or compliance with the study procedures
* Participants with current hepatitis A virus (HAV) infection (confirmed by HAV antibody immunoglobulin M [IgM]), hepatitis A virus (HBV) infection (confirmed by hepatitis A virus [HBsAg]), and hepatitis C virus (HCV) infection (confirmed by HCV antibody) at screening. Evidence of clinically relevant active infection that would interfere with study conduct or its interpretation is also exclusionary
* Participants with current human immunodeficiency virus (HIV) type 1 (HIV-1) or type 2 (HIV-2) infection (confirmed by antibodies) at screening
* Male participants with pregnant partners
* Male participants who plan to father a child while enrolled in this study or within 90 days after the last dose of study drug
* Participants who have taken any disallowed therapies as noted in Prohibitions and Restrictions Section, and Concomitant Medications Section, before the planned first dose of study drug
* Participants having used immune-modulating agents within 6 months prior the first dosing of study drugs, for example, immunosuppressants, interferon alpha (IFN-alpha), or oral corticosteroids
* Participants having received an investigational agent or investigational vaccine or used an invasive investigational medical device within 12 weeks, or having received a biological product within 12 weeks or 5 half-lives (whichever is longer) prior to the first dosing of study drugs
* Participants participating in another clinical or medical interventional research study
* Participants with a) Greater than or equal to (>=) Grade 1 laboratory abnormalities at screening as defined by the Division of Acquired Immune Deficiency Syndrome (DAIDS) Toxicity Grading Scale; or b) Total bilirubin outside the normal range Note: Retesting of abnormal laboratory values that may lead to exclusion will be allowed once without prior asking approval from the Sponsor. Retesting will take place during an unscheduled visit in the screening phase. Participants with a normal value at retest may be included
* Participants who had major surgery (for example, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study, or within 12 weeks after the last dose of study drug Note: Participants with planned surgical procedures to be conducted under local anesthesia may participate
* Participant is an employee of the Sponsor, the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the investigator NOTE: Investigators should ensure that all study enrollment criteria have been met at screening. If a participant's clinical status changes (including any available laboratory results or receipt of additional medical records) after screening but before the first dose of study drug is given or before the follow-up period, such that he or she no longer meets all eligibility criteria, then the participant should be excluded from participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately up to 9 weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Part 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately up to 12 weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Part 1: Number of Participants With AEs by Severity | Approximately up to 9 weeks
  Severity of AEs will be graded according to the Division of Acquired Immune Deficiency Syndrome (DAIDS) Toxicity Grading Scale as follows: Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe); Grade 4 (potentially life-threatening); and Grade 5 (death related to the AE).
Part 2: Number of Participants With AEs by Severity | Approximately up to 12 weeks
  Severity of AEs will be graded according to the Division of AIDS (DAIDS) Toxicity Grading Scale as follows: Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe); Grade 4 (potentially life-threatening); and Grade 5 (death related to the AE).
Part 1: Number of Participants with Clinically Significant Changes in Physical Examination | Approximately up to 9 weeks
  Number of participants with clinically significant changes in the physical examination (including height, body weight measurement, and skin examination) will be reported.
Part 2: Number of Participants with Clinically Significant Changes in Physical Examination | Approximately up to 12 weeks
  Number of participants with clinically significant changes in the physical examination (including height, body weight measurement, and skin examination) will be reported.
Part 1: Number of Participants with Vital Sign Abnormalities | Approximately up to 9 weeks
  Number of participants with vital signs abnormalities (vital signs includes body temperature, pulse rate, respiratory rate, oxygen saturation [SaO2] and blood pressure) will be reported.
Part 2: Number of Participants with Vital Sign Abnormalities | Approximately up to 12 weeks
  Number of participants with vital signs abnormalities (vital signs includes body temperature, pulse rate, respiratory rate, oxygen saturation [SaO2] and blood pressure) will be reported.
Part 1: Number of Participants with Laboratory Abnormalities | Approximately up to 9 weeks
  Number of participants with clinical laboratory abnormalities (serum chemistry, hematology, and coagulation) will be reported.
Part 2: Number of Participants with Laboratory Abnormalities | Approximately up to 12 weeks
  Number of participants with clinical laboratory abnormalities (serum chemistry, hematology, and coagulation) will be reported.
Part 1: Number of Participants with Holter Monitoring Abnormalities | Approximately up to 9 weeks
  Number of participants with Holter monitoring abnormalities (related to heart's activity such as rate and rhythm) will be reported.
Part 2: Number of Participants with Holter Monitoring Abnormalities | Approximately up to 12 weeks
  Number of participants with Holter monitoring abnormalities (related to heart's activity such as rate and rhythm) will be reported.
Part 1: Number of Participants with Electrocardiogram (ECG) Abnormalities | Approximately up to 9 weeks
  Number of participants with electrocardiogram (ECG) abnormalities will be reported.
Part 2: Number of Participants with Electrocardiogram (ECG) Abnormalities | Approximately up to 12 weeks
  Number of participants with electrocardiogram (ECG) abnormalities will be reported.
Part 1: Number of Participants with Cytokine Release Syndrome (CRS) | Approximately up to 9 weeks
  Number of participants with CRS will be reported. CRS is defined as a disorder characterized by nausea, headache, tachycardia, hypotension, rash, and/or shortness of breath.
Part 2: Number of Participants with Cytokine Release Syndrome (CRS) | Approximately up to 12 weeks
  Number of participants with CRS will be reported. CRS is defined as a disorder characterized by nausea, headache, tachycardia, hypotension, rash, and/or shortness of breath.
Part 1: Number of Participants with Cytokine Release Syndrome (CRS) by Severity | Approximately up to 9 weeks
  Severity of CRS will be graded according to DAIDS as follows: Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe); and Grade 4 (potentially life-threatening).
Part 2: Number of Participants with Cytokine Release Syndrome (CRS) by Severity | Approximately up to 12 weeks
  Severity of CRS will be graded according to DAIDS as follows: Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe); and Grade 4 (potentially life-threatening).
Part 1: Maximum Observed Plasma Concentration (Cmax) of AL-034 Following Single Dose Administration in Fasted State | Day 1: predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose
  The Cmax is the maximum observed concentration of AL-034 in plasma following single ascending dose (SAD) administration.
Part 2: Maximum Observed Plasma Concentration (Cmax) of AL-034 Following Repeated Dose Administration | Days 1, 22, and 29: predose, and 0.5, 1, 2, and 12 hours postdose
  The Cmax is the maximum observed concentration of AL-034 in plasma following multiple ascending dose (MAD) administration.
Part 1: Area Under the Plasma Concentration Time Curve (AUC) of AL-034 Following Single Dose Administration in Fasted State | Day 1: predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose
  AUC is the area under the plasma concentration time curve of AL-034 in plasma following SAD administration.
Part 2: Area Under the Plasma Concentration Time Curve (AUC) of AL-034 Following Repeated Dose Administration | Days 1, 22, and 29: predose, and 0.5, 1, 2, and 12 hours postdose
  AUC is the area under the plasma concentration time curve of AL-034 in plasma following MAD administration.
Part 1: AL-034 Concentration in Urine Following a Single Dose Administration | Day 1: 0 to 6, 6 to 12, and 12 to 24 hours postdose
  Concentration in urine of AL-034 following a single dose administration will be determined.
Part 2: AL-034 Concentration in Urine Following Repeated Dose Administration | Day 1: 0 to 6, 6 to 12, and 12 to 24 hours postdose
  Concentration in urine of AL-034 following MAD administration will be determined.

SECONDARY OUTCOMES:
Part 1: Maximum Observed Plasma Concentration (Cmax) of AL-034 Following Single Dose Administration in Fed State | Day 1: predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose
  The Cmax is the maximum observed concentration of AL-034 in plasma following SAD administration.
Part 2: Area Under the Plasma Concentration Time Curve (AUC) of AL-034 Following Single Dose Administration in Fed State | Day 1: predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose
  AUC is the area under the plasma concentration time curve of AL-034 in plasma following SAD administration.

CONTACTS AND LOCATIONS:
Overall Officials: Alios Biopharma Inc. Clinical Trial, Study Director — Alios Biopharma Inc.
Locations (1):
- Auckland Clinical Studies, Ltd., Auckland, New Zealand

REFERENCES:
- [Background] Bazett HC. An analysis of the time-relationship of electrocardiograms. Heart. 1920; 7:353 380.
- [Background] Di Bisceglie AM. Hepatitis B and hepatocellular carcinoma. Hepatology. 2009 May;49(5 Suppl):S56-60. doi: 10.1002/hep.22962. PMID 19399807
- [Background] Chang TT, Gish RG, de Man R, Gadano A, Sollano J, Chao YC, Lok AS, Han KH, Goodman Z, Zhu J, Cross A, DeHertogh D, Wilber R, Colonno R, Apelian D; BEHoLD AI463022 Study Group. A comparison of entecavir and lamivudine for HBeAg-positive chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1001-10. doi: 10.1056/NEJMoa051285. PMID 16525137
- [Background] Cohen C, Holmberg SD, McMahon BJ, Block JM, Brosgart CL, Gish RG, London WT, Block TM. Is chronic hepatitis B being undertreated in the United States? J Viral Hepat. 2011 Jun;18(6):377-83. doi: 10.1111/j.1365-2893.2010.01401.x. Epub 2010 Dec 8. PMID 21143343
- [Background] European Association For The Study Of The Liver. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012 Jul;57(1):167-85. doi: 10.1016/j.jhep.2012.02.010. Epub 2012 Mar 20. No abstract available. PMID 22436845
- [Background] Fridericia LS. Die Systolendauer im Elektrokardiogramm bei normalen Menschen und bei Herzkranken. Acta Med Scand 1920; 53: 469-486
- [Background] Investigator's Brochure: JNJ 64794964 (AL-034). Edition 1. Janssen Research & Development (May 2017).
- [Background] Lai CL, Shouval D, Lok AS, Chang TT, Cheinquer H, Goodman Z, DeHertogh D, Wilber R, Zink RC, Cross A, Colonno R, Fernandes L; BEHoLD AI463027 Study Group. Entecavir versus lamivudine for patients with HBeAg-negative chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1011-20. doi: 10.1056/NEJMoa051287. PMID 16525138
- [Background] Liang TJ. Hepatitis B: the virus and disease. Hepatology. 2009 May;49(5 Suppl):S13-21. doi: 10.1002/hep.22881. PMID 19399811
- [Background] Lok AS, McMahon BJ, Brown RS Jr, Wong JB, Ahmed AT, Farah W, Almasri J, Alahdab F, Benkhadra K, Mouchli MA, Singh S, Mohamed EA, Abu Dabrh AM, Prokop LJ, Wang Z, Murad MH, Mohammed K. Antiviral therapy for chronic hepatitis B viral infection in adults: A systematic review and meta-analysis. Hepatology. 2016 Jan;63(1):284-306. doi: 10.1002/hep.28280. Epub 2015 Nov 13. PMID 26566246
- [Background] Lucifora J, Protzer U. Attacking hepatitis B virus cccDNA--The holy grail to hepatitis B cure. J Hepatol. 2016 Apr;64(1 Suppl):S41-S48. doi: 10.1016/j.jhep.2016.02.009. PMID 27084036
- [Background] Marcellin P, Lau GK, Bonino F, Farci P, Hadziyannis S, Jin R, Lu ZM, Piratvisuth T, Germanidis G, Yurdaydin C, Diago M, Gurel S, Lai MY, Button P, Pluck N; Peginterferon Alfa-2a HBeAg-Negative Chronic Hepatitis B Study Group. Peginterferon alfa-2a alone, lamivudine alone, and the two in combination in patients with HBeAg-negative chronic hepatitis B. N Engl J Med. 2004 Sep 16;351(12):1206-17. doi: 10.1056/NEJMoa040431. PMID 15371578
- [Background] Phyo WW, Soh AY, Lim SG, Lee GH. Search for a cure for chronic hepatitis B infection: How close are we? World J Hepatol. 2015 May 28;7(9):1272-81. doi: 10.4254/wjh.v7.i9.1272. PMID 26019743
- [Background] Poggio ED, Wang X, Greene T, Van Lente F, Hall PM. Performance of the modification of diet in renal disease and Cockcroft-Gault equations in the estimation of GFR in health and in chronic kidney disease. J Am Soc Nephrol. 2005 Feb;16(2):459-66. doi: 10.1681/ASN.2004060447. Epub 2004 Dec 22. PMID 15615823
- [Background] Schweitzer A, Horn J, Mikolajczyk RT, Krause G, Ott JJ. Estimations of worldwide prevalence of chronic hepatitis B virus infection: a systematic review of data published between 1965 and 2013. Lancet. 2015 Oct 17;386(10003):1546-55. doi: 10.1016/S0140-6736(15)61412-X. Epub 2015 Jul 28. PMID 26231459
- [Background] Williamson DF. Descriptive epidemiology of body weight and weight change in U.S. adults. Ann Intern Med. 1993 Oct 1;119(7 Pt 2):646-9. doi: 10.7326/0003-4819-119-7_part_2-199310011-00004. PMID 8363190
- [Background] World Health Organization (WHO). Hepatitis B Fact Sheet. Available at: http://www.who.int/mediacentre/factsheets/fs204/en/. Accessed 31 January 2017